CLINICAL TRIAL: NCT04206735
Title: Implementation of Interprofessional Training to Improve Uptake of Noninvasive Ventilation in Patients Hospitalized With Severe COPD Exacerbation
Brief Title: The Impact of Interprofessional Training to Improve the Uptake of Noninvasive Ventilation in Patients Hospitalized With Severe COPD Exacerbation
Acronym: COPD-NIV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Complications to recruiting due to COVID-19 pandemic
Sponsor: Baystate Medical Center (Other)
Collaborators: University of Illinois at Chicago (Other); University of North Carolina, Chapel Hill (Other); Premier Inc (Industry); Tufts Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1351436; R01HL146615 (NIH)
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Copd
Keywords: Interprofessional training; Education; Noninvasive ventilation; Mechanical ventilation; Non-randomized open cohort step-wedge
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Hospitals that agree to participate are offered 3 dates at approximately 6-month intervals. They sign up for a date depending on their readiness to participate. A team of champions: nurses, respiratory therapists (RTs), and physicians from each hospital will attend a virtual one-day training which will include NIV knowledge, skills, and the principles of teamwork. The clinicians in the participating institutions will be then on how to appropriately deliver NIV know and the principles of teamwork by an online course and by the champions teams.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interprofessional Education (IPE) (Experimental): Each hospital needs to assign a 'COPD-NIV' team of champions to lead the implementation strategy at the local level. We will provide virtual or in-person (if safety permits) training for the COPD-NIV teams (one RT, one RN, and one MD). The training will consist of NIV knowledge and skills through the principles of IPE and teamwork. We will use the train the trainer method; after we train the COPD-NIV team champions, the champions will promote and hold training sessions for their peers in person (if safety permits, 2-3 times a month for 4 months). At present, we are providing these training sessions as prerecorded content available whenever the clinician is available. Champions will promote the training to their clinicians for the first 4 months and then at 6 and 12 months for new staff.
  Interventions: Other: Interprofessional Education (IPE); Other: Usual care

INTERVENTIONS:
Other: Interprofessional Education (IPE) — We will use the training stated in the arm description above. In addition, prerecorded webinars that include evidence-based practice management of COPD will be released every month for the champions and clinicians to watch at their leisure.
Other: Usual care — Usual care of patients hospitalized with severe COPD exacerbation

SUMMARY:
COPD is the fourth leading cause of death in the US, and COPD exacerbations result in approximately 700,000 hospitalizations annually. Patients who do not respond to pharmacotherapy are placed on invasive (IMV) or noninvasive mechanical ventilation (NIV). Studies have shown that patients treated with NIV are less likely to require IMV and have better mortality and length of hospital stay. NIV is recommended in COPD guidelines as the first-line of treatment for patients with severe exacerbation who have failed pharmacologic treatment. Yet, despite compelling evidence of benefit, there is substantial variation in the implementation of NIV across hospitals, leading to preventable morbidity and mortality. The main goal of this project is to determine the impact of inter-professional educational strategies in 20 hospitals with low NIV use in COPD by using a non-randomized stepped-wedge open cohort design. Inter-professional education (IPE) targets complex team-based care in NIV delivery. The central hypothesis is that inter-professional education on how to care for patients with COPD using NIV will lead to improvement in the uptake of NIV, and that respiratory therapist (RT autonomy) and team functionality will act as mediators.

DETAILED DESCRIPTION:
COPD is the fourth leading cause of death in the US, and COPD exacerbations result in approximately 700,000 hospitalizations annually. Patients who do not respond to pharmacotherapy are placed on invasive mechanical ventilation (IMV) or noninvasive mechanical ventilation (NIV). Although IMV reverses hypercapnia/hypoxia, it can cause significant morbidity and mortality. NIV is an alternative ventilatory option for acute respiratory failure that provides positive pressure ventilation via a mask. Multiple randomized controlled trials and analyses of real-world data have shown that patients treated with NIV are less likely to require IMV, and have lower mortality and length of hospital stay. NIV is recommended in COPD guidelines as the first-line treatment for patients with severe exacerbation who have failed pharmacologic treatment. Yet, despite compelling evidence of benefit, we have previously demonstrated substantial variation in the implementation of NIV across hospitals, leading to preventable morbidity and mortality.

Through a series of mixed-methods studies, we have found that successful implementation of NIV requires physicians, respiratory therapists (RTs), and nurses to communicate and collaborate effectively to select appropriate patients for treatment, and to carefully manage patients after NIV initiation. These studies suggest that efforts to increase the use of NIV in COPD need to account for the complex and interdisciplinary nature of NIV delivery and the need for team coordination. The main goal of this project is to determine the impact of interprofessional educational (IPE) strategies in 20 hospitals with low NIV use in COPD by conducting non-randomized open cohort step wedge trial. The IPE will target complex team-based care in NIV delivery. The primary outcome of the trial is change in the hospital rate of NIV use among patients with COPD requiring ventilatory support. The central hypothesis is that IPE will lead to improvement in the uptake of NIV, and that RT autonomy and team functionality will act as mediators. The goal will be accomplished by completing three specific aims. Aim 1 will compare the change in NIV use over time among patients with COPD in hospitals enrolled by comparing their NIV rates from before the IPE training, to after the training. Aim 2 will explore mediators' role (RT autonomy and team functionality) on the relationship between the implementation strategies and implementation effectiveness. In Aim 3, we will assess the acceptability and feasibility of the educational training through interviews with providers. This proposal is significant because NIV is the only therapy that has been shown to improve short-term survival for patients hospitalized for exacerbation of COPD, yet a large number of hospitals still have not adopted this approach fully.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitals with low rates of NIV use (lower-half quartiles) among patients with COPD ventilated with invasive or noninvasive mechanical ventilation. Rates are calculated from an administrative database. Hospitals must also have a minimum of 10 ventilated patients over an 18 month period per hospital in which to assess NIV rates. (the above age limits are for patients with COPD included in calculating the rates)
2. The target population of clinicians for the IPE educational training aged 23-80 years includes: physicians (hospitalists, emergency department physicians, critical care or pulmonary), respiratory therapists, and nurses involved in the care of patients with COPD or acute respiratory failure at the participating hospitals.

Exclusion Criteria:

None

Ages: 23 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-08 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Changes in the use of NIV | At baseline and 18 months after baseline
  Hospitals' rate of NIV among ventilated COPD patients at 18 and 36 months
Sustainability | 36 months after training is completed
  Hospitals' rate of NIV among ventilated COPD patients/Administrative database.If there are no changes in NIV among ventilated patients after 18 months then we will not examine sustainability of the training at 36 months after training is completed.
Acceptability and feasibility of the educational training | At 18 months after baseline
  Interviews with providers will be conducted to determine the acceptability and feasibility of the educational training
Penenetration of training | 18 months after training is completed
  Proportion of providers completing the training (assessed using participation logs)
Changes in Respiratory Therapist Job Autonomy | Pre-training (baseline), 12 months after training, 36 months after training
  Survey of RTs regarding their belief on how autonomous they are in delivering NIV
Changes in team functionality | Pre-training (baseline), 12 months after training, 36 months after training
  Survey of physicians, RTs and nurses regarding team functionality in delivering NIV

SECONDARY OUTCOMES:
Changes in NIV failure rates | Pre-training (baseline), 12 months after training, 36 months after training
  Hospitals' rate of NIV failure among all COPD patients
Changes in hospital length of stay | Pre-training (baseline), 12 months after training, 36 months after training
  Median Hospital length of stay among all COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Stefan, Phd. MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center (Institute for Healthcare and Population Science), Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
7. The dataset submitted to NHLBI will be prepared in accordance with the requirements for NHLBI data repository datasets and associated documentation for submission and the NHLBI Policy for Data Sharing for Clinical Trials and Epidemiological Studies, and in accordance with the Guidelines for NHLBI Data Set Preparation
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: one year after the study completion
Access Criteria: By request from investigators. The protocol will be published

REFERENCES:
- [Background] Stefan MS, Pekow PS, Shieh MS, Hill NS, Rothberg MB, Fisher KA, Lindenauer PK. Hospital Volume and Outcomes of Noninvasive Ventilation in Patients Hospitalized With an Acute Exacerbation of Chronic Obstructive Pulmonary Disease. Crit Care Med. 2017 Jan;45(1):20-27. doi: 10.1097/CCM.0000000000002006. PMID 27509388
- [Background] Stefan MS, Shieh MS, Pekow PS, Hill N, Rothberg MB, Lindenauer PK. Trends in mechanical ventilation among patients hospitalized with acute exacerbations of COPD in the United States, 2001 to 2011. Chest. 2015 Apr;147(4):959-968. doi: 10.1378/chest.14-1216. PMID 25375230
- [Background] Lindenauer PK, Stefan MS, Shieh MS, Pekow PS, Rothberg MB, Hill NS. Outcomes associated with invasive and noninvasive ventilation among patients hospitalized with exacerbations of chronic obstructive pulmonary disease. JAMA Intern Med. 2014 Dec;174(12):1982-93. doi: 10.1001/jamainternmed.2014.5430. PMID 25347545
- [Background] Fisher KA, Mazor KM, Goff S, Stefan MS, Pekow PS, Williams LA, Rastegar V, Rothberg MB, Hill NS, Lindenauer PK. Successful Use of Noninvasive Ventilation in Chronic Obstructive Pulmonary Disease. How Do High-Performing Hospitals Do It? Ann Am Thorac Soc. 2017 Nov;14(11):1674-1681. doi: 10.1513/AnnalsATS.201612-1005OC. PMID 28719228
- [Background] Hughes AM, Gregory ME, Joseph DL, Sonesh SC, Marlow SL, Lacerenza CN, Benishek LE, King HB, Salas E. Saving lives: A meta-analysis of team training in healthcare. J Appl Psychol. 2016 Sep;101(9):1266-304. doi: 10.1037/apl0000120. Epub 2016 Jun 16. PMID 27599089
- [Background] Marlow SL, Hughes AM, Sonesh SC, Gregory ME, Lacerenza CN, Benishek LE, Woods AL, Hernandez C, Salas E. A Systematic Review of Team Training in Health Care: Ten Questions. Jt Comm J Qual Patient Saf. 2017 Apr;43(4):197-204. doi: 10.1016/j.jcjq.2016.12.004. Epub 2017 Feb 16. PMID 28325208
- [Background] Stefan MS, Nathanson BH, Higgins TL, Steingrub JS, Lagu T, Rothberg MB, Lindenauer PK. Comparative Effectiveness of Noninvasive and Invasive Ventilation in Critically Ill Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease. Crit Care Med. 2015 Jul;43(7):1386-94. doi: 10.1097/CCM.0000000000000945. PMID 25768682
- [Background] Metcalf AY, Stoller JK, Habermann M, Fry TD. Respiratory Therapist Job Perceptions: The Impact of Protocol Use. Respir Care. 2015 Nov;60(11):1556-9. doi: 10.4187/respcare.04156. Epub 2015 Aug 25. PMID 26306735
- [Derived] Stefan MS, Pekow PS, Shea CM, Hughes AM, Hill NS, Steingrub JS, Farmer MJS, Hess DR, Riska KL, Clark TA, Lindenauer PK. Update to the study protocol for an implementation-effectiveness trial comparing two education strategies for improving the uptake of noninvasive ventilation in patients with severe COPD exacerbation. Trials. 2021 Dec 16;22(1):926. doi: 10.1186/s13063-021-05855-9. PMID 34915905
- [Derived] Stefan MS, Pekow PS, Shea CM, Hughes AM, Hill NS, Steingrub JS, Lindenauer PK. Protocol for two-arm pragmatic cluster randomized hybrid implementation-effectiveness trial comparing two education strategies for improving the uptake of noninvasive ventilation in patients with severe COPD exacerbation. Implement Sci Commun. 2020;1(1):46. doi: 10.1186/s43058-020-00028-2. Epub 2020 May 6. PMID 32435762